CLINICAL TRIAL: NCT02181673
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Trial of Golimumab, an Anti-TNFα Monoclonal Antibody, Administered Intravenously, in Subjects With Active Psoriatic Arthritis
Brief Title: A Study of Golimumab in Participants With Active Psoriatic Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR103796; 2014-000242-30 (EudraCT Number); CNTO148PSA3001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2014-07-02; First posted 2014-07-04 (Estimated); Results first posted 2017-12-21 (Actual); Last update posted 2017-12-21 (Actual); Status verified 2017-12

CONDITIONS: Arthritis, Psoriatic
Keywords: Psoriatic arthritis; Golimumab; Simponi
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — golimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Group 1: Placebo (Placebo Comparator): Participants will receive intravenous infusions of placebo at Weeks 0, 4, 12 and 20. At Week 24, all participants receiving placebo will begin receiving intravenous infusions of golimumab 2 milligram per kilogram (mg/kg) at Week 24, 28 and thereafter every 8 weeks up to Week 52.
  Interventions: Drug: Placebo; Drug: Golimumab
- Treatment Group 2: Golimumab (Experimental): Participants will receive intravenous infusions of golimumab 2 mg/kg at Weeks 0, 4 and thereafter every 8 weeks up to Week 52. At Week 24, participants will receive a placebo infusion to maintain the blind.
  Interventions: Drug: Placebo; Drug: Golimumab

INTERVENTIONS:
Drug: Placebo — Participants will receive intravenous infusions of placebo at Weeks 0, 4, 12 and 20 in treatment Group 1 and intravenous infusions of placebo at Week 24 to maintain the blind in treatment Group 2.
Drug: Golimumab — Participants will receive intravenous infusions of golimumab 2mg/kg at Weeks 0, 4 and thereafter every 8 weeks up to Week 52 in treatment Group 2 and intravenous infusions of golimumab (2mg/kg) at Weeks 24, 28 and thereafter every 8 weeks up to Week 52 in treatment Group 1.

SUMMARY:
The purpose of this study is to evaluate the efficacy of intravenously (administration of a fluid into the vein) administered golimumab 2 milligram per kilogram (mg/kg) in participants with active psoriatic arthritis (a chronic inflammatory arthritis that is associated with psoriasis).

DETAILED DESCRIPTION:
This is a Phase 3, multicenter (when more than one hospital or medical school team work on a medical research study), randomized (study drug assigned by chance), double-blind (neither the researchers nor the participants know what treatment the participant is receiving), placebo-controlled (an inactive substance; a pretend treatment [with no drug in it] that is compared in a clinical trial with a drug to test if the drug has a real effect) study of golimumab compared with placebo in participants with active psoriatic arthritis. The study will include 4 phases: Screening phase (up to 6 weeks), Double-blind placebo-controlled phase (Week 0 to Week 24), Active treatment phase (Week 24 to Week 52), and Safety follow-up phase (8 weeks from last study drug administration). Total duration of the study will be 60 weeks per participant. Eligible Participants will be randomly assigned to either Treatment Group 1: Placebo or Treatment Group 2: Golimumab. Participants randomized to Placebo Group, will receive intravenous infusions of placebo at Weeks 0, 4, 12 and 20. At Week 24, all participants receiving placebo will begin receiving intravenous infusions of golimumab (2 mg/kg) at Week 24, 28 and thereafter every 8 weeks up to Week 52. Participants randomized to Golimumab Group, will receive intravenous infusions of golimumab 2 mg/kg at Week 0, 4 and thereafter every 8 weeks up to Week 52. At Week 24, participants randomized to golimumab Group will receive a placebo infusion to maintain the blind. The efficacy will be assessed primarily by measuring percentage of participants who achieve a 20 percent improvement from baseline in the assessment used in active psoriatic arthritis at Week 14. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Have had psoriatic arthritis (PsA) for at least 6 months prior to the first administration of study agent
* Have a diagnosis of active PSA as defined by 5 or more swollen joints and 5 or more tender joints at Screening and at Baseline and C-reactive protein >=0.6 milligram per deciliter (mg/dL) at Screening
* Have active plaque psoriasis or a documented history of plaque psoriasis
* Have active PsA despite current or previous disease-modifying antirheumatic drugs (DMARD) and/or nonsteroidal anti-inflammatory drug (NSAID) therapy. DMARD therapy is defined as taking a DMARD for at least 3 months, or evidence of DMARD intolerance. NSAID therapy is defined as taking an NSAID for at least 4 weeks or evidence of NSAID intolerance

Exclusion Criteria:

* Have other inflammatory diseases that might confound the evaluations of benefit of Golimumab therapy, including but not limited to rheumatoid arthritis, ankylosing spondylitis, systemic lupus erythematosus, or Lyme disease
* Are pregnant, nursing, or planning a pregnancy or fathering a child while enrolled in the study or within 4 months after receiving the last administration of study agent
* Have used any biologic agents that are targeted for reducing tumor necrosis factors (TNF) alpha, including but not limited to Infliximab, Etanercept, Adalimumab, Golimumab, and Certolizumab Pegol
* Have ever used cytotoxic drugs, including Chlorambucil, Cyclophosphamide, Nitrogen mustard, or other Alkylating agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2014-09-08 (Actual); Primary Completion 2016-05-05 (Actual); Study Completion 2017-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (88):
- United States (13):
  - Glendale, Arizona
  - Mesa, Arizona
  - Huntington Beach, California
  - Lakewood, California
  - Granger, Indiana
  - Indianapolis, Indiana
  - Monroe, Louisiana
  - Tupelo, Mississippi
  - St Louis, Missouri
  - Orchard Park, New York
  - Salisbury, North Carolina
  - Duncansville, Pennsylvania
  - Austin, Texas
- Australia (2):
  - Daw Park
  - Maroochydore
- Belarus (4):
  - Grodno
  - Homyel
  - Minsk
  - Vitebsk
- Canada (3):
  - St. John's, Newfoundland and Labrador
  - Waterloo, Ontario
  - Burlington
- Germany (7):
  - Bad Doberan
  - Berlin
  - Cologne
  - Erfurt
  - Hamburg
  - Ratingen
  - Zerbst
- Hungary (7):
  - Balatonfüred
  - Budapest
  - Debrecen
  - Hévíz
  - Kistarcsa
  - Nyíregyháza
  - Szombathely
- Lithuania (5):
  - Alytus
  - Kaunas
  - Klaipėda
  - Šiauliai
  - Vilnius
- Poland (10):
  - Bydgoszcz
  - Bytom
  - Częstochowa
  - Krakow
  - Lublin
  - Nadarzyn
  - Nowa Sól
  - Poznan
  - Warsaw
  - Wroclaw
- Romania (4):
  - Bucharest
  - Constanța
  - Iași
  - Ploieşti
- Russia (16):
  - Kemerovo
  - Korolyov
  - Krasnoyarsk
  - Kursk
  - Moscow
  - Novosibirsk
  - Orenburg
  - Petrozavodsk
  - Ryazan
  - Saint Petersburg
  - Saratov
  - Tomsk
  - Tver'
  - Ulyanovsk
  - Vladimir
  - Yaroslavl
- Spain (3):
  - Córdoba
  - Getafe
  - Seville
- Ukraine (14):
  - Chernihiv
  - Dnipropetrovsk
  - Kharkiv
  - Khmelnitsky
  - Kryvyi Rih
  - Kyiv
  - Lviv
  - Odesa
  - Poltava
  - Sumy
  - Ternopil
  - Uzhhorod
  - Vinnytsia
  - Zaporizhzhia

REFERENCES:
- [Derived] Husni ME, Deodhar A, Schwartzman S, Chakravarty SD, Hsia EC, Leu JH, Zhou Y, Lo KH, Kavanaugh A. Pooled safety results across phase 3 randomized trials of intravenous golimumab in rheumatoid arthritis, psoriatic arthritis, and ankylosing spondylitis. Arthritis Res Ther. 2022 Mar 21;24(1):73. doi: 10.1186/s13075-022-02753-6. PMID 35313978
- [Derived] Mease P, Husni ME, Kafka S, Chakravarty SD, Harrison DD, Lo KH, Xu S, Hsia EC, Kavanaugh A. Inhibition of radiographic progression across levels of composite index-defined disease activity in patients with active psoriatic arthritis treated with intravenous golimumab: results from a phase-3, double-blind, placebo-controlled trial. Arthritis Res Ther. 2020 Mar 6;22(1):43. doi: 10.1186/s13075-020-2126-1. PMID 32143685
- [Derived] Husni ME, Kavanaugh A, Murphy F, Rekalov D, Harrison DD, Kim L, Lo KH, Leu JH, Hsia EC. Efficacy and Safety of Intravenous Golimumab Through One Year in Patients With Active Psoriatic Arthritis. Arthritis Care Res (Hoboken). 2020 Jun;72(6):806-813. doi: 10.1002/acr.23905. Epub 2020 May 15. PMID 30980514
- [Derived] Kavanaugh A, Husni ME, Harrison DD, Kim L, Lo KH, Noonan L, Hsia EC. Radiographic Progression Inhibition with Intravenous Golimumab in Psoriatic Arthritis: Week 24 Results of a Phase III, Randomized, Double-blind, Placebo-controlled Trial. J Rheumatol. 2019 Jun;46(6):595-602. doi: 10.3899/jrheum.180681. Epub 2019 Feb 15. PMID 30770519
- [Derived] Kavanaugh A, Husni ME, Harrison DD, Kim L, Lo KH, Leu JH, Hsia EC. Safety and Efficacy of Intravenous Golimumab in Patients With Active Psoriatic Arthritis: Results Through Week Twenty-Four of the GO-VIBRANT Study. Arthritis Rheumatol. 2017 Nov;69(11):2151-2161. doi: 10.1002/art.40226. PMID 28805045

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo (Week 0-24): Participants received intravenous infusions of placebo at Weeks 0, 4, 12 and 20.
- Placebo Then Golimumab 2 mg/kg (Week 24-60): Participants who received placebo up to Week 20 were then crossed over at Week 24 to receive intravenous infusions of golimumab 2 milligram per kilogram (mg/kg) at Week 24, 28 and every 8 weeks thereafter up to Week 52.
- Golimumab 2 mg/kg (Week 0-60): Participants were randomized to receive intravenous infusions of golimumab 2 mg/kg at Weeks 0, 4 and every 8 weeks thereafter up to Week 52. At Week 24, participants received a placebo intravenous infusion to maintain the blind.
Period: Up to Week 24
Arm/Group | Placebo (Week 0-24) | Placebo Then Golimumab 2 mg/kg (Week 24-60) | Golimumab 2 mg/kg (Week 0-60)
Started | 239 | 0 | 241
Treated | 239 | 0 | 240
Completed | 222 | 0 | 230
Not Completed | 17 | 0 | 11
Not completed — Adverse Event | 2 | 0 | 3
Not completed — Death | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 3
Not completed — Withdrawal by Subject | 10 | 0 | 1
Not completed — Other | 2 | 0 | 3
Not completed — Randomized not Treated | 0 | 0 | 1
Period: Week 24-Week 60
Arm/Group | Placebo (Week 0-24) | Placebo Then Golimumab 2 mg/kg (Week 24-60) | Golimumab 2 mg/kg (Week 0-60)
Started | 0 | 222 | 230
Treated | 0 | 220 | 230
Completed | 0 | 214 | 213
Not Completed | 0 | 8 | 17
Not completed — Adverse Event | 0 | 4 | 10
Not completed — Other | 0 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 2
Not completed — Pregnancy | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Golimumab 2 mg/kg: Participants were randomized to receive intravenous infusions of golimumab 2 mg/kg at Weeks 0, 4 and every 8 weeks thereafter up to Week 52. At Week 24, participants received a placebo intravenous infusion to maintain the blind.
- Total: Total of all reporting groups
Arm/Group | Placebo (Week 0-24) | Golimumab 2 mg/kg | Total
Number analyzed (Participants) | 239 | 241 | 480
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 0 | 2
  Between 18 and 65 years | 216 | 228 | 444
  >=65 years | 21 | 13 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (12.53) | 45.7 (11.25) | 46.2 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 113 | 231
  Male | 121 | 128 | 249
Region of Enrollment [Count of Participants; unit: Participants]
  Belarus | 14 | 8 | 22
  Canada | 1 | 0 | 1
  Germany | 3 | 1 | 4
  Hungary | 13 | 9 | 22
  Lithuania | 13 | 17 | 30
  Poland | 43 | 34 | 77
  Romania | 3 | 1 | 4
  Russian Federation | 79 | 74 | 153
  Spain | 1 | 2 | 3
  Ukraine | 61 | 86 | 147
  United States | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved an American College of Rheumatology (ACR) 20 Response at Week 14
Description: The ACR 20 response is defined as greater than or equal to (>=) 20 percent (%) improvement from baseline in both swollen joint count (66 joints) and tender joint count (68 joints) and >=20% improvement from baseline in at least 3 of the following 5 assessments: Patient's assessment of pain (on a 0 to 10 centimeter [cm] scale), Patient's Global Assessment of Disease Activity (on a 0 to 10 cm scale), Physician's Global Assessment of Disease Activity (on a 0 to 10 cm scale), Patient's assessment of physical function as measured by Disability Index of the Health Assessment Questionnaire (HAQ-DI) and measurement of a blood test called C-reactive protein (CRP).
Time Frame: Week 14
Population: The full analysis set (FAS) included all participants who were randomized.
Measure: Number; unit: Percentage of Participants
Groups:
- Placebo: Participants received intravenous infusions of placebo at Weeks 0, 4, 12 and 20.
- Golimumab: Participants were randomized to receive intravenous infusions of golimumab 2 mg/kg at Weeks 0, 4 and thereafter every 8 weeks up to Week 52. At Week 24, participants received a placebo infusion to maintain the blind.
Arm/Group | Placebo | Golimumab
Number analyzed (Participants) | 239 | 241
Percentage of Participants | 21.8 | 75.1
Statistical Analysis 1: Comparison: Placebo vs Golimumab; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Percent Difference = 53.4, 95% CI 2-sided [45.80 to 60.90]

2. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at Week 14
Description: The Health Assessment Questionnaire-Disability Index (HAQ-DI) is a 20-question instrument that assesses the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping and activities of daily living). Responses in each functional area are scored from 0 to 3 (0=no difficulty and 3=inability to perform a task in that area). Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty.
Time Frame: Baseline and Week 14
Population: The full analysis set (FAS) included all participants who were randomized. Here "N" (number of participants analyzed) signifies the number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Golimumab
Number analyzed (Participants) | 222 | 233
units on a scale | -0.12 (0.466) | -0.60 (0.530)

3. Secondary Outcome: Percentage of Participants Who Achieved an ACR 50 Response at Week 14
Description: The ACR 50 response is defined as: greater than or equal to (>=) 50 percent (%) improvement from baseline in both swollen joint count (66 joints) and tender joint count (68 joints) and >=50% improvement from baseline in at least 3 of the following 5 assessments: Patient's assessment of pain (on a 0 to 10 cm scale), Patient's Global Assessment of Disease Activity (on a 0 to 10 cm scale), Physician's Global Assessment of Disease Activity (on a 0 to 10 cm scale), Patient's assessment of physical function as measured by Disability Index of the Health Assessment Questionnaire (HAQ-DI) and measurement of a blood test called C-reactive protein (CRP).
Time Frame: Week 14
Population: The full analysis set (FAS) included all participants who were randomized.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Golimumab
Number analyzed (Participants) | 239 | 241
Percentage of Participants | 6.3 | 43.6

4. Secondary Outcome: Percentage of Participants Who Achieved Psoriatic Area and Severity Index (PASI) 75 Response at Week 14
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas were assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 to 6, and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease. A PASI 75 response represents participants who achieved at least a 75 percent improvement from baseline in the PASI score.
Time Frame: Week 14
Population: The analysis set included randomized participants with greater than or equal to (>=) 3 percent (%) body surface area (BSA) Psoriasis Skin Involvement at Baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Golimumab
Number analyzed (Participants) | 198 | 196
Percentage of participants | 13.6 | 59.2

5. Secondary Outcome: Change From Baseline in Total Modified Van Der Heijde-Sharp (vdH-S) Score at Week 24
Description: The modified vdH-S score is a radiographic evaluation of hand and feet erosions and joint space narrowing (JSN) for 20 joints per hand and 6 joints per foot with a total score ranging from 0 (best) to 528 (worst = worst possible erosion score of 320 + worst possible JSN score of 208). Higher score and positive score changes indicate more radiographic damage and radiographic progression, respectively.
Time Frame: Baseline and Week 24
Population: FAS for structural damage endpoints (FAS-SD) defined as participants in the FAS who were treated and had a non-missing baseline total modified vdH-S score for the analysis.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Golimumab
Number analyzed (Participants) | 237 | 237
units on a scale | 1.95 (0.264) | -0.36 (0.144)

6. Secondary Outcome: Change From Baseline in Leeds Enthesitis Index (LEI) at Week 14 in Participants With Enthesitis at Baseline
Description: Enthesitis will be assessed using the Leeds Enthesitis Index (LEI). The LEI was developed to assess enthesitis in participants with PsA, and evaluates the presence (score of 1) or absence of pain (score of 0) by applying local pressure to Lateral elbow epicondyle, left and right, Medial femoral condyle, left and right, and Achilles tendon insertion, left and right. LEI scores ranging from 0 (0 sites with tenderness) to 6 (worst possible score; 6 sites with tenderness).
Time Frame: Baseline and Week 14
Population: Population included all randomized participants with Enthesitis at Baseline. Here "N" (number of participants analyzed) signifies the number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Golimumab
Number analyzed (Participants) | 173 | 182
units on a scale | -0.8 (1.98) | -1.8 (1.75)

7. Secondary Outcome: Change From Baseline in Dactylitis Scores at Week 14 in Participants With Dactylitis at Baseline
Description: Dactylitis is characterized by swelling of the entire finger or toe. The severity of dactylitis is scored on a scale of 0-3, where 0=tenderness and 3=extreme tenderness in each digit of the hands and feet. The range of total dactylitis scores for a participant is 0-60. Higher score indicates greater degree of tenderness.
Time Frame: Baseline and Week 14
Population: Population included all Randomized participants With Dactylitis (Score >0) at Baseline. Here "N" (number of participants analyzed) signifies the number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Golimumab
Number analyzed (Participants) | 115 | 130
units on a scale | -2.8 (7.03) | -7.8 (8.57)

8. Secondary Outcome: Change From Baseline in Short Form-36 Health Survey (SF-36) Physical Component Summary (PCS) at Week 14
Description: The SF-36 is a survey of participant health. It consists of 8 individual domains, which are weighted sums of the questions in their section. The 8 domains are: vitality (VT), physical functioning (PF), bodily pain (BP), general health (GH), Role-Physical (RP), Role-Emotional (RE), social functioning (SF) and mental health (MH). Each of these 8 scales (domains) is scored from 0 to 100 with higher scores indicating better health. Based on the scale scores, the summary physical component score (PCS) is derived. Scales contributing most to the scoring of the SF-36 PCS include the PF, RP, BP and GH. Other domains not noted contribute to the scoring but to a lesser degree. The scoring is derived based on an algorithm that has been developed in a software provided by the developer. The summary PCS score is also scaled from 0 to 100 with higher scores indicating better health.
Time Frame: Baseline and Week 14
Population: The full analysis set (FAS) included all participants who were randomized. Here "N" (number of participants analyzed) signifies the number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Golimumab
Number analyzed (Participants) | 222 | 233
units on a scale | 2.69 (5.920) | 8.65 (7.602)

9. Secondary Outcome: Percentage of Participants Who Achieved an American College of Rheumatology (ACR) 50 Response at Week 24
Description: The ACR 50 response is defined as greater than or equal to (>=) 50 percent (%) improvement from baseline in both swollen joint count (66 joints) and tender joint count (68 joints) and >=50% improvement from baseline in at least 3 of the following 5 assessments: Patient's assessment of pain (on a 0 to 10 centimeter [cm] scale), Patient's Global Assessment of Disease Activity (on a 0 to 10 cm scale), Physician's Global Assessment of Disease Activity (on a 0 to 10 cm scale), Patient's assessment of physical function as measured by Disability Index of the Health Assessment Questionnaire (HAQ-DI) and measurement of a blood test called C-reactive protein (CRP).
Time Frame: Week 24
Population: The full analysis set (FAS) included all participants who were randomized.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Golimumab
Number analyzed (Participants) | 239 | 241
Percentage of participants | 6.3 | 53.5

10. Secondary Outcome: Percentage of Participants Who Achieved an American College of Rheumatology (ACR) 70 Response at Week 14
Description: The ACR 70 response is defined as greater than or equal to (>=) 70 percent (%) improvement from baseline in both swollen joint count (66 joints) and tender joint count (68 joints) and >=70% improvement from baseline in at least 3 of the following 5 assessments: Patient's assessment of pain (on a 0 to 10 centimeter [cm] scale), Patient's Global Assessment of Disease Activity (on a 0 to 10 cm scale), Physician's Global Assessment of Disease Activity (on a 0 to 10 cm scale), Patient's assessment of physical function as measured by Disability Index of the Health Assessment Questionnaire (HAQ-DI) and measurement of a blood test called C-reactive protein (CRP).
Time Frame: Week 14
Population: The full analysis set (FAS) included all participants who were randomized.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Golimumab
Number analyzed (Participants) | 239 | 241
Percentage of participants | 2.1 | 24.5

11. Secondary Outcome: Change From Baseline in Short Form-36 Health Survey (SF)-36 Mental Component Summary (MCS) at Week 14
Description: The SF-36 is a survey of participant health. It consists of 8 individual domains, which are weighted sums of the questions in their section. The 8 domains are: vitality (VT), physical functioning (PF), bodily pain (BP), general health (GH), Role-Physical (RP), Role-Emotional (RE), social functioning (SF) and mental health (MH). Each of these 8 scales (domains) is scored from 0 to 100 with higher scores indicating better health. Based on the scale scores, the summary mental component score (MCS) is derived. Scales contributing most to the scoring of the SF-36 MCS include the VT, SF, RE and MH. Other domains not noted contribute to the scoring but to a lesser degree. The scoring is derived based on an algorithm that has been developed in a software provided by the developer. The summary MCS score is also scaled from 0 to 100 with higher scores indicating better health.
Time Frame: Baseline and Week 14
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Golimumab
Number analyzed (Participants) | 222 | 233
units on a scale | 0.97 (7.644) | 5.33 (9.948)

ADVERSE EVENTS:
Time Frame: Up to 60 Weeks
Description: Safety Population included all participants who received at least 1 dose of study agent.
Arm/Group | Placebo (Week 0-24) | Placebo Then Golimumab 2 mg/kg (Week 24-60) | Golimumab 2 mg/kg (Week 0-60)
Serious Adverse Events (participants affected / at risk) | 8/239 | 5/220 | 19/240
Other Adverse Events (participants affected / at risk) | 19/239 | 25/220 | 40/240
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Week 0-24) (N=239) | Placebo Then Golimumab 2 mg/kg (Week 24-60) (N=220) | Golimumab 2 mg/kg (Week 0-60) (N=240)
Cardiac failure acute (Cardiac disorders) | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 1 | 0 | 0
Oedematous pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Hepatitis chronic active (Hepatobiliary disorders) | 0 | 0 | 1
Empyema (Infections and infestations) | 0 | 1 | 0
Infected dermal cyst (Infections and infestations) | 0 | 0 | 1
Periodontitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 2
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 2
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Epidural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Gene mutation identification test positive (Investigations) | 0 | 1 | 0
Laboratory test abnormal (Investigations) | 0 | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pleomorphic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebral haematoma (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1
Neuritis (Nervous system disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Week 0-24) (N=239) | Placebo Then Golimumab 2 mg/kg (Week 24-60) (N=220) | Golimumab 2 mg/kg (Week 0-60) (N=240)
Nasopharyngitis (Infections and infestations) | 13 | 9 | 14
Alanine aminotransferase increased (Investigations) | 5 | 13 | 25
Aspartate aminotransferase increased (Investigations) | 5 | 12 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.